CLINICAL TRIAL: NCT06412666
Title: A Phase 2/3 Multicenter, Randomized, Double-Blind, Placebo-Controlled and Open-Label Extension Trial to Evaluate the Efficacy and Safety of Aficamten in a Pediatric Population With Symptomatic Obstructive Hypertrophic Cardiomyopathy
Brief Title: A Study to Evaluate the Effect of Aficamten in Pediatric Patients With Symptomatic Obstructive Hypertrophic Cardiomyopathy (oHCM).
Acronym: CEDAR-HCM
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CY 6023; 2024-511377-30-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-05

CONDITIONS: Pediatric; Symptomatic Obstructive Hypertrophic Cardiomyopathy
Keywords: CK-3773274; CK-274; Aficamten; Symptomatic Obstructive Hypertrophic Cardiomyopathy; oHCM; CEDAR; CEDAR-HCM; CY 6023

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aficamten (Experimental): Participants in this arm will receive a single daily oral dose of aficamten with dose levels (5 mg to 20 mg) guided by echocardiography assessments, for 12 weeks during the double-blinded period, for another 52 weeks during the open-label extension period, and for an additional 144 weeks during the long-term extension period.
  Interventions: Drug: Aficamten
- Placebo (Placebo Comparator): Participants in this arm will receive a single daily oral dose of placebo for 12 weeks during the double-blinded period and then will receive aficamten for 52 weeks during the open-label extension period, followed by an additional 144 weeks of aficamten during the long-term extension period.
  Interventions: Drug: Aficamten; Drug: Placebo

INTERVENTIONS:
Drug: Aficamten — Oral Tablet
Drug: Placebo — Oral Tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and PK of aficamten in a pediatric population with symptomatic obstructive hypertrophic cardiomyopathy (oHCM).

DETAILED DESCRIPTION:
The overall objective of the trial is to determine the efficacy, safety, and tolerability of administration of aficamten in adolescents (12 to < 18 years old) and children (6 to < 12 years old) with symptomatic oHCM. Adolescents and children will be studied in a staged approach involving established favorable pharmacodynamic and safety profiles of aficamten in adolescents followed by further pharmacokinetic modeling to inform the dosing regimen in children. Only the 12 to <18 years old cohort is currently open for enrollment.

The trial will consist of 3 periods:

1. Period 1 is the randomized, double-blind, placebo-controlled treatment period that will assess the efficacy, safety and tolerability of aficamten in pediatric participants. Duration: 12 weeks.
2. Period 2 is the open-label extension trial that will assess the long-term safety of aficamten in pediatric participants, and further assess efficacy and tolerability. Duration: 52 weeks.
3. Period 3 is the long-term extension trial that will assess the long-term safety of aficamten in pediatric participants, and further assess efficacy and tolerability. Duration: 144 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Period 1: Treatment Period

  * Males and females between 12 and < 18 years of age at screening and at Day 1.
  * Body weight ≥ 45 kg for the initial cohort and then body weight ≥ 35 kg after at least 10 participants in the initial cohort have undergone dose titration up to Week 4 without observed events of LVEF < 50% at the starting dose of 5 mg qd.
  * Core laboratory confirmation of the following oHCM echocardiographic criteria at screening:
* Left ventricular (LV) hypertrophy with nondilated LV chamber in the absence of other cardiac disease.
* LV end-diastolic wall thickness that meets a threshold of:

  * Z-score > 2.5 in the absence of family history OR
  * Z-score > 2 in the presence of positive family history or positive genetic test.
* LVEF ≥ 60% AND Valsalva LVOT-G ≥ 50 mmHg.

  * oHCM of sarcomeric origin confirmed by genetic testing or, if unable to confirm by genetic testing, oHCM of sarcomeric origin may be presumed in the absence of history of metabolic disorders, mitochondrial cardiomyopathies, neuromuscular disease, malformation syndromes, infiltrative diseases/inflammation, and endocrine disorders (such as Fabry's disease, Noonan syndrome with left ventricular hypertrophy, and amyloid-cardiomyopathy).
  * New York Heart Association (NYHA) Class ≥ II at screening.
  * Adequate acoustic windows for echocardiography.
  * Participants on beta blockers, verapamil, diltiazem, or disopyramide should have been on stable doses for more than 4 weeks prior to randomization.
* Period 2: Open-Label Extension

  * Completed Period 1. If unable to complete Period 1 due to circumstances not related to compliance or safety, the Medical Monitor may review and determine eligibility.
  * LVEF ≥ 55% after washout.
* Period 3: Long-term Extension • Completed Period 2.

Exclusion Criteria:

* Period 1: Treatment Period

Any of the following criteria will exclude potential participants from the trial:

* Significant valvular heart disease.

  * Moderate or severe valvular aortic stenosis or fixed subaortic obstruction.
  * Mitral regurgitation that is greater than mild in severity and not due to systolic anterior motion of the mitral valve (per judgment of Principal Investigator or designee).
  * Evidence of fixed left-sided obstruction (eg, subaortic membrane, aortic valve stenosis, or coarctation of the aorta).
* History of LV systolic dysfunction (LVEF < 45%) or stress cardiomyopathy at any time during their clinical course.
* History of congenital heart disease other than oHCM (may be enrolled if not hemodynamically significant in the judgement of the Principal Investigator and study Medical Monitor).
* Has been treated with SRT (surgical myectomy or percutaneous alcohol septal ablation) within the preceding 6 months or has plans for either treatment during the trial period.
* History of paroxysmal or persistent atrial fibrillation or atrial flutter.
* History of syncope, symptomatic ventricular arrhythmia, or sustained ventricular tachyarrhythmia within 3 months prior to screening.
* History or evidence of any other clinically significant disorder, malignancy, active infection, other condition, or disease that, in the opinion of the Principal Investigator (or designee) or the Medical Monitor, would pose a risk to participant safety or interfere with the trial evaluation, procedures, or completion.
* Current or previous use of drugs known to cause cardiomyopathy (eg, anthracyclines, monoclonal antibodies [trastuzumab], alkylating agents [cyclophosphamide], and tyrosine kinase inhibitors [sunitinib and imatinib]).
* Currently participating in another investigational device or drug trial or received an investigational device or drug < 1 month (or 5 half-lives for drugs, whichever is longer) prior to screening.
* Implantable cardioverter defibrillator (ICD) implantation within 6 weeks of screening or planned ICD implantation during the trial period.
* Has received prior treatment with aficamten or mavacamten.
* Currently listed for heart transplantation or anticipated to be listed for heart transplantation in the next 12 months.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Valsalva left ventricular outflow tract gradient (LVOT-G) | Baseline to week 12

SECONDARY OUTCOMES:
Change from baseline in resting LVOT-G | Baseline to week 12
Change in values of NT-proBNP | Baseline to week 12
Change in values of hs-cTnI | Baseline to week 12
Change in New York Heart Association (NYHA) Functional Class | Baseline to week 12
Proportion of patients with ≥1 class improvement in NYHA Functional Class | Baseline to week 12
Trough observed plasma concentration (Ctrough) and C2h postdose of aficamten | Baseline to week 12
Maximum observed concentration (Cmax), tmax, AUCtau, and Ctrough of aficamten | Week 8 or Week 12
  A voluntary intensive PK substudy may occur at Week 8 or Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Cytokinetics MD, Study Director — Cytokinetics
Locations (38):
- United States (26):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Hospital, Washington D.C., District of Columbia
  - Nicklaus Children's Hospital, Miami, Florida
  - Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Morristown Medical Center, Morristown, New Jersey
  - NYP/Columbia University Medical Center, New York, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Duke Clinical Research Institute, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - LeBonheur Children's Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Dell Children's Hospital, Austin, Texas
  - UT Southwestern, Dallas, Texas
  - Children's Wisconsin, Milwaukee, Wisconsin
- The Hospital for Sick Children (SickKids), Toronto, Ontario, Canada
- Careggi University Hospital, Florence, Italy
- Japan (5):
  - NHO Kagoshima Medical Center, Kagoshima
  - University of Osaka Hospital, Osaka
  - Kitasato University Hospital, Sagamihara
  - National Cerebral and Cardiovascular Center, Suita
  - Juntendo University Hospital, Tokyo
- Spain (2):
  - Unidad de Cardiología Infantil; Hospital Universitario da Coruña, A Coruña
  - Hospital Sant Joan de Deu, Barcelona
- United Kingdom (3):
  - Alder Hey Children's Hospital, Liverpool
  - Evelina Children's Hospital, London
  - Great Ormond Street Hospital for Children, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaski JP, Kantor PF, Nakano SJ, Olivotto I, Russell MW, Godown J, Chiu M, German P, Heitner SB, Jacoby DL, Kupfer S, Lutz J, Maharao N, Malik FI, Melloni C, Nieto Morales PF, Simkins T, Wei J, Ho CY; CEDAR-HCM Investigators. Efficacy and Safety of Aficamten in Children and Adolescents With Obstructive Hypertrophic Cardiomyopathy: Study Design and Rationale of CEDAR-HCM. Circ Heart Fail. 2025 Dec 5:e013418. doi: 10.1161/CIRCHEARTFAILURE.125.013418. Online ahead of print. PMID 41347307